CLINICAL TRIAL: NCT03411889
Title: A Study to Develop a Protocol for Functional Magnetic Resonance Imaging of the Lacrimal Drainage System
Brief Title: A Feasibility Study to Develop a Protocol for Functional Lacrimal Magnetic Resonance Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 225255
Record Dates: First submitted 2018-01-04; First posted 2018-01-26 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Lacrimal Duct Obstruction; Lacrimal Stenosis
MeSH Terms: conditions — Lacrimal Duct Obstruction | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- functional lacrimal delay (Experimental): Participants shown to have functional delay on DSG will be included. The intervention will be an MRI scan during tear drainage
  Interventions: Diagnostic Test: MRI scanning

INTERVENTIONS:
Diagnostic Test: MRI scanning — MRI scanning during tear drainage
  Other Names: functional MRI

SUMMARY:
Watering eyes (epiphora) is a very common ophthalmic condition. It is frequently caused by dysfunction of the lacrimal (tear) drainage system which is the 'pipework' that takes tears from the eye to the nasal cavity. If the system is completely blocked then the patient is offered surgery to unblock or bypass the obstruction. However, the system is often either partially obstructed, or there is tear drainage delay despite there being no apparent obstruction (functional obstruction). Currently this is investigated with two separate scans, conducted at different times in different departments (CT and nuclear medicine). These are dacryocystography (DCG) and dacryoscintigraphy (DSG) and both are required as they have different limitations and benefits. Moreover DCG is a CT scan that uses radiation.

Functional magnetic resonance dacryocystography (MR DCG) is increasingly widely used in other fields of medicine (e.g. cardiology) because of the increasing acquisition speed and resolution of MRI scanners in recent years. The investigators anticipate functional MRI of the lacrimal drainage system (i.e. scanning as eye drops are instilled and pass down the system) will overcome the shortcomings of DCG and DSG, by simultaneously providing both good anatomical detail and physiological images. Various methods of MR DCG have been described in the literature and there is no standard protocol for this procedure as of current. In this study, the investigators aim to develop a protocol for MR DCG that can be used in routine radiological practice in place of DCG and DSG and get pilot data on tear drainage in participants with known delayed tear drainage and controls with normal tear drainage systems.

DETAILED DESCRIPTION:
Tear drainage delay is a common problem that causes a watery eye. This can impair activities of daily living such as reading and driving, can be a huge nuisance requiring continual dabbing with a tissue and can cause infections and abscesses of the tear drainage system. The current, standard investigations for tear drainage delay have significant limitations with two separate scans in separate departments being required. A functional MRI scan would be able to combine these two scans and provide both better anatomical and functional detail than each one respectively. This would have several major benefits:

1. Improved diagnostic information to guide the treatment choice
2. Reduced scan resource usage as one scan would provide all the required functional anatomical and functional information.
3. Improved patient convenience
4. Improved safety as radiation is used for CT DCG, where MRI The study involves investigation of both controls with normal tear drainage and individuals with known tear drainage delay. Both groups are required for the development of the protocol as the speed of tear transit will differ greatly which will facilitate optimisation of the MRI scan protocol. This will also provide preliminary data on the speed of tear passage in a normal lacrimal drainage system and in an impaired system.

Several other functional lacrimal drainage MRI studies have been done. However, a clear protocol has not been developed and there is no data on normal and abnormal MRI appearances and tear transit times.

The normal standard of care will not be delayed by this investigation as it will be conducted while patients are awaiting other lacrimal investigations (DCG and DSG) or lacrimal surgery, none of which would be affected by this study.

ELIGIBILITY:
Inclusion Criteria:

* Lacrimal drainage disease participants (n=5)

  1. Symptomatic epiphora (tearing)
  2. Nasolacrimal drainage dysfunction confirmed by the following characteristics:

     1. An abnormal delay of tear transit on DSG
     2. A normal DCG and lacrimal syringing investigation
     3. Normal eyelid and punctal anatomy

Controls

1. No epiphora
2. Normal lacrimal syringing in clinic.

Exclusion criteria

1. Age under 18
2. Renal function <30mL/min/1.73m2
3. Contra-indications to MRI e.g. electronic or metal implants, severe claustrophobia
4. Known adverse reactions to contrast agents
5. Pregnancy

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
A protocol for functional MRI scanning | 60 minutes. This is a feasibility study in which participants are seen on one occasion and have one MRI scan which is expected to take around 60 minutes
  This is a feasibility study for functional MRI scanning. The primary outcome is a MRI scanning protocol that can be routinely used to assess the 'real-time' drainage of lacrimal flow

CONTACTS AND LOCATIONS:
Locations (1):
- Brighton & Sussex University Hospitals, Brighton, East Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No